CLINICAL TRIAL: NCT07069764
Title: Efficacy of Photobiomodulation Therapy Using 980nm Versus 635nm Diode Lasers for Treatment of Myofascial Pain
Acronym: LLLTsEMG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Laser Enhanced Sciences (Other)
Responsible Party: Principal Investigator, Dr. Hala Shaaban, Dentist, National Institute of Laser Enhanced Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NILES-TMD-LLLT-2024; TMD-NILES-STUDY-LASER-TRIAL-20 (Other: NILES, Cairo University)
Record Dates: First submitted 2025-07-07; First posted 2025-07-17 (Actual); Results first posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-09

CONDITIONS: Myofascial Pain Syndrome
Keywords: Low-Level Laser Therapy
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Intervention Model Description: "Randomized controlled trial with two parallel groups comparing the effect of low-level diode laser therapy at 980 nm and 635 nm wavelengths on myofascial pain in temporomandibular disorders. Participants receive treatment sessions over a defined period with outcomes measured by surface electromyography and pain scales."
Masking Description: "This is an open-label study with no masking; both participants and investigators are aware of the treatment assignments."
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-Level Laser Therapy at 635 nm for Arm 1 (Experimental): Participants will receive low-level laser therapy using a diode laser with 635 nm wavelength, applied 2 times per week for 5 weeks to treat myofascial pain syndrome in the temporomandibular joint.
  Interventions: Device: Doctor smile 635nm For Arm 1
- Low-Level Laser Therapy at 980 nm for Arm 2 (Experimental): Participants will receive low-level laser therapy using a diode laser with 980 nm wavelength, applied 2 times per week for 5 weeks to treat myofascial pain syndrome in the temporomandibular joint.
  Interventions: Device: Doctor smile 980 nm For Arm2

INTERVENTIONS:
Device: Doctor smile 635nm For Arm 1 — Participants will receive low-level laser therapy using a diode laser with a wavelength of 635 nanometers. The treatment will be applied twice weekly for five weeks to the affected temporomandibular joint muscles to reduce myofascial pain and improve muscle function.
  Other Names: device_LLLT
  Arms: Low-Level Laser Therapy at 635 nm for Arm 1
Device: Doctor smile 980 nm For Arm2 — Participants will receive low-level laser therapy using a diode laser with a wavelength of 980 nanometers. The treatment will be applied twice weekly for five weeks to the affected temporomandibular joint muscles to reduce myofascial pain and improve muscle function.
  Other Names: device _LLLT
  Arms: Low-Level Laser Therapy at 980 nm for Arm 2

SUMMARY:
This randomized controlled clinical trial aims to evaluate the efficacy of low-level laser therapy (LLLT) using two different diode laser wavelengths (980 nm and 635 nm) in the treatment of myofascial pain associated with temporomandibular disorders (TMD). The study compares pain reduction and muscle activity improvement using surface electromyography (sEMG) before and after laser application. Participants are randomly assigned to receive either 980 nm or 635 nm laser treatment twice per week for five weeks. The primary outcomes include pain intensity and functional mandibular movements, while secondary outcomes assess changes in sEMG recordings.

DETAILED DESCRIPTION:
This randomized controlled clinical trial investigates the effectiveness of low-level laser therapy (LLLT) using two diode laser wavelengths-980 nm and 635 nm-for the treatment of myofascial pain syndrome (MPS) in patients with temporomandibular disorders (TMD). The study is conducted at the National Institute of Laser Enhanced Sciences (NILES), Cairo University.

Participants who meet the inclusion criteria are randomly assigned to two intervention groups. Group 1 receives LLLT using a 635 nm diode laser, while Group 2 receives LLLT using a 980 nm diode laser. Both groups undergo treatment twice per week for a total of five weeks, following a standardized protocol.

The primary outcomes include pain intensity assessed using a visual analog scale (VAS), and evaluation of mandibular range of motion including lateral and protrusive movements. Secondary outcomes involve the assessment of masseter and temporalis muscle activity using surface electromyography (sEMG) before and after the treatment period.

The study aims to provide evidence-based comparison between the two wavelengths in terms of pain reduction and neuromuscular improvement, contributing to the optimization of non-invasive laser protocols for TMD-related myofascial pain.

ELIGIBILITY:
Inclusion Criteria:

* - patients with myofascial pain due to stress, medically free, not to resort to self-medication during the study period with no chronic diseases.

Exclusion Criteria:

* Patients with TMJ disorders either due to bony degeneration changes or soft tissue changes.
* Patients with pain of dental etiology were excluded, pregnancy, lactation, cardiac arrhythmia, diabetic patients, erosions and medically free.
* Patient with history of malignancy or a history of previous surgery of neck and/ shoulder within the past year of the study were excluded.
* Any patients had treatment that can affect muscles will be excluded, either pharmacological treatment (e.g, opioids, morphine, muscles relaxants or anti-depressants), physiotherapy management and occlusal splints.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — "Eligible for both male and female participants
Enrollment: 30 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-03-29 (Actual); Study Completion 2025-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: hala SH Attiyah, BDS, Principal Investigator — National Institute of Laser Enhanced Sciences (NILES), Cairo University
Locations (1):
- National Institute for Laser Enhanced Sciences, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the data will be used only within the study team for internal analysis, and no external data sharing is planned.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low-Level Laser Therapy at 635 nm for Arm 1 | Low-Level Laser Therapy at 980 nm for Arm 2
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants (15 in each group) were included in the baseline analysis population.
Groups:
- Low-Level Laser Therapy at 635 nm for Arm 1: Participants received low-level laser therapy using a diode laser with a 635 nm wavelength. Treatment was applied twice weekly for five weeks to the masticatory muscles affected by myofascial pain syndrome in the temporomandibular joint region, aiming to reduce pain and improve muscle function.
- Low-Level Laser Therapy at 980 nm for Arm 2: Participants received low-level laser therapy using a diode laser with 980 nm wavelength, applied 2 times per week for 5 weeks to treat myofascial pain syndrome in the temporomandibular joint.
  Doctor smile 980 nm For Arm2: Participants will receive low-level laser therapy using a diode laser with a wavelength of 980 nanometers. The treatment will be applied twice weekly for five weeks to the affected temporomandibular joint muscles to reduce myofascial pain and improve muscle function.
- Total: Total of all reporting groups
Arm/Group | Low-Level Laser Therapy at 635 nm for Arm 1 | Low-Level Laser Therapy at 980 nm for Arm 2 | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] — "Participant age range at baseline was 18 to 50 years
  years | 29.6 (6.5) | 30.1 (7) | 29.9 (6.7)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Distribution of participants by sex at baseline.
  Participants
    male | 7 | 8 | 15
    female | 8 | 7 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants] — Distribution of participants by race/ethnicity was assessed at baseline according to NIH/OMB standard categories.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 15 | 15 | 30
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Distribution of participants by race/ethnicity was assessed at baseline according to NIH/OMB standard categories.
  Participants
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 15 | 15 | 30
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity Reduction
Description: "Pain intensity was assessed in patients with myofascial pain syndrome of the temporomandibular joint using the Visual Analog Scale (VAS), a 10-point scale ranging from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate greater pain intensity. Measurements were recorded at baseline, after 10 sessions of low-level laser therapy (5 weeks), and at 1-month follow-up. Data are reported in the tables below. Lower scores reflect reduced pain intensity
Time Frame: At baseline, after 10 treatment sessions (5 weeks), and at 1-month follow-up (approximately 2 months in total from baseline).
Population: "All randomized participants in each arm (15 participants per group) were included in the analysis population. Analyses were conducted according to the intention-to-treat principle, including all participants who received at least one session of low-level laser therapy and had at least one post-baseline assessment."
Measure: Mean (Standard Deviation); unit: "units on scale
Arm/Group | Low-Level Laser Therapy at 635 nm for Arm 1 | Low-Level Laser Therapy at 980 nm for Arm 2
Number analyzed (Participants) | 15 | 15
"units on scale
  Baseline | 7.6 (1.2) | 7.8 (1.1)
  Post-treatment(after 10 sessions) | 3.2 (1.1) | 2.5 (1.0)
  AFTER one month | 2.9 (1.3) | 2.1 (0.9)
Statistical Analysis 1: Comparison: Low-Level Laser Therapy at 635 nm for Arm 1 vs Low-Level Laser Therapy at 980 nm for Arm 2; "The study was designed to compare the effects of 635 nm and 980 nm low-level laser therapy on pain and jaw function. Statistical analysis methods are described below."; Test type: Other — "This study was not designed as a non-inferiority or equivalence trial. It was powered (80% power, α = 0.05) to detect clinically significant differences in pain reduction between 635 nm and 980 nm diode lasers, based on prior LLLT studies in TMD. Sample size was calculated before recruitment."; p = 0.05, Friedman test, Mann-Whitney U test — P-values were adjusted using Bonferroni correction for multiple comparisons. The a priori threshold for statistical significance was set at p < 0.05; Non-parametric tests were used due to non-normal data distribution (Shapiro-Wilk test). Effect size measures were also reported; Effect size (Kendall's W and r) = 0.75, 95% CI 2-sided [0.68 to 0.79]; "Shapiro-Wilk test was used to assess normality. Non-parametric tests were applied. Friedman test for within-group comparisons, followed by Bonferroni-adjusted post hoc tests. Mann-Whitney U test for between-group comparisons. Effect sizes were calculated using Kendall's W (within groups) and r (between groups)."

2. Secondary Outcome: Maximum Mouth Opening (MMO)
Description: "Maximum Mouth Opening (MMO) was assessed in millimeters at three time points: baseline, after 10 sessions of low-level laser therapy (5 weeks), and at 1-month follow-up. Data are reported as mean ± standard deviation in the tables below. No conclusions or comparisons are included in this description."
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Low-Level Laser Therapy at 635 nm for Arm 1 | Low-Level Laser Therapy at 980 nm for Arm 2
Number analyzed (Participants) | 15 | 15
millimeters
  baseline | 34.5 (4.2) | 34 (3.9)
  after 10 sessions | 41.3 (3.5) | 43.5 (3.2)
  follow up after 1 month | 42.1 (3.2) | 44.2 (2.9)

3. Secondary Outcome: Lateral Jaw Movements
Description: Lateral jaw movements (side-to-side excursion) were measured in millimeters to assess changes in temporomandibular joint function. Measurements were recorded at baseline, after 10 sessions of low-level laser therapy (5 weeks), and at 1-month follow-up. Higher values indicate a greater range of mandibular motion.
Time Frame: as for outcome 1
Population: All randomized participants completed the study and were included in the analysis for this outcome measure.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Low-Level Laser Therapy at 635 nm for Arm 1 | Low-Level Laser Therapy at 980 nm for Arm 2
Number analyzed (Participants) | 15 | 15
millimeters
  baseline | 6.2 (0.9) | 6.0 (0.8)
  after 10 sessions | 8.3 (1.0) | 8.7 (1.1)
  follow up after one month | 8.5 (0.8) | 8.8 (1)

4. Secondary Outcome: Changes in Muscle Activity Measured by Surface Electromyography (sEMG)
Description: Surface electromyography (sEMG) was used to assess the electrical activity of the masseter and anterior temporalis muscles during maximum voluntary clenching. Recordings were obtained at baseline and after 10 sessions of low-level laser therapy (5 weeks). Results are expressed as mean amplitude values in microvolts (µV). Lower values indicate reduced muscle activity, which reflects clinical improvement.
Time Frame: At baseline and after 10 treatment sessions (5 weeks)
Population: sEMG analysis includes participants with valid baseline and post-treatment data. Differences in numbers are due to technical issues, poor signal quality, or withdrawals. Variations in sample size reflect missing data for some muscles or time points
Measure: Mean (Standard Deviation); unit: microvolts
Groups:
- Low-Level Laser Therapy at 980 nm for Arm 2: Participants treated with 980 nm low-level laser therapy; muscle activity was measured by surface electromyography (sEMG) before and after treatment sessions.
- Low-Level Laser Therapy at 635 nm for Arm 1: Participants treated with 635 nm low-level laser therapy; muscle activity was measured by surface electromyography (sEMG) before and after treatment sessions.
Arm/Group | Low-Level Laser Therapy at 980 nm for Arm 2 | Low-Level Laser Therapy at 635 nm for Arm 1
Number analyzed (Participants) | 15 | 15
microvolts
  Right temporalis M before treatment | 15.8 (2.9) | 15.5 (3.1)
  Right temporalis M after 10 sessions | 8.9 (2.3) | 9.9 (2.9)
  Left temporalis M before treatment | 16.1 (3.0) | 15.9 (3)
  Left temporalis M after 10 sessions | 9.2 (2.4) | 10.1 (2.8)
  Right masster M before treatment | 16.8 (2.9) | 16.5 (3.1)
  Right masseter M after 10 sessions | 8.9 (2.3) | 9.9 (2.9)
  Left masseter M before treatment | 17.2 (3.3) | 16.8 (3.2)
  Left masseter M after 10 sessions | 8.5 (2.2) | 10.2 (2.7)

5. Secondary Outcome: Protrusive Movements
Description: Protrusive mandibular movements were measured in millimeters to evaluate the functional improvement of the temporomandibular joint. Measurements were taken at baseline, after 5 weeks of low-level laser therapy, and at 1-month follow-up. Higher values indicate greater range of mandibular protrusive motion.
Time Frame: as for outcome 1
Population: randomized participants who completed the study protocol were included in the analysis. No participants were excluded from the outcome measure analysis."
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Low-Level Laser Therapy at 635 nm for Arm 1 | Low-Level Laser Therapy at 980 nm for Arm 2
Number analyzed (Participants) | 15 | 15
millimeters
  baseline | 5.8 (0.7) | 5.9 (0.6)
  after 10 sessions | 7.4 (0.8) | 7.8 (0.7)
  follow up after one month | 7.5 (0.7) | 8.0 (0.6)

ADVERSE EVENTS:
Time Frame: "Adverse event data were collected from baseline, throughout the 5-week treatment period, and at the 1-month follow-up visit."
Description: "The standard definitions of adverse events and serious adverse events, as provided by ClinicalTrials.gov, were used. Data were collected systematically through patient self-reports and clinical observations during treatment sessions and at the follow-up visit."
Groups:
- Low-Level Laser Therapy at 635 nm for Arm 1: Participants received photobiomodulation therapy using a diode laser at a wavelength of 635 nm. Treatment was applied twice per week for 5 weeks to the masseter and temporalis muscles associated with temporomandibular disorder. The goal was to reduce myofascial pain and improve mandibular function.
- Low-Level Laser Therapy at 980 nm for Arm 2: Participants received photobiomodulation therapy using a diode laser at a wavelength of 980 nm. Treatment was applied twice per week for 5 weeks to the masseter and temporalis muscles associated with temporomandibular disorder. The goal was to reduce myofascial pain and improve mandibular function.
Arm/Group | Low-Level Laser Therapy at 635 nm for Arm 1 | Low-Level Laser Therapy at 980 nm for Arm 2
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-Level Laser Therapy at 635 nm for Arm 1 (N=15) | Low-Level Laser Therapy at 980 nm for Arm 2 (N=15)
No adverse events reported (Eye disorders) | 0 (0) | 0 (0) — "No ocular adverse effects reported due to the use of protective eye goggles during laser therapy
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-Level Laser Therapy at 635 nm for Arm 1 (N=15) | Low-Level Laser Therapy at 980 nm for Arm 2 (N=15)
None reported (General disorders) | 0 (0) | 0 (0) — No adverse events or side effects were observed or reported by participants during or after the low-level laser therapy treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-03-25): https://cdn.clinicaltrials.gov/large-docs/64/NCT07069764/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/64/NCT07069764/SAP_001.pdf